CLINICAL TRIAL: NCT02839447
Title: A Clinical Evaluation of Semen Quality Using the MiOXSYS™ System 2.0
Status: Withdrawn | Type: Observational
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Aytu BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PCL-0002
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Male Infertility
Keywords: semen; sperm; oxidative stress; reactive oxygen species; idiopathic male infertility
MeSH Terms: conditions — Infertility, Male | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human male semen containing sperm
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Semen: Semen that meet the criteria for "normal" on sperm number, motility, and morphology as described by the current WHO manual.
  Interventions: Diagnostic Test: Diagnostic
- Abnormal Semen: Semen that fail to achieve one or more of the criteria for "normal" on sperm number, motility, and morphology as described by the current WHO manual.
  Interventions: Diagnostic Test: Diagnostic

INTERVENTIONS:
Diagnostic Test: Diagnostic — Diagnostic

SUMMARY:
The purpose of this study is to determine if elevations in oxidative stress, as measured by oxidation-reduction potential (ORP), can distinguish between semen samples from men with abnormal semen parameters from those with normal semen parameters. Static ORP (sORP) results, measured by the MiOXSYS System- a novel technology, will be compared to the current World Health Organization (WHO) semen analysis parameters (5th Edition WHO Laboratory Manual for the Examination and Processing of Human Semen [2010]).

DETAILED DESCRIPTION:
Oxidative stress reflects an imbalance in the redox system in favor of the activity of reactive oxygen species and other free radicals. It is also dependent upon the biological system's ability to detoxify these oxidative compounds through the application of antioxidants and other reductants. Disturbances in the normal redox state can cause adverse effects on cells including protein oxidation, lipid peroxidation, and DNA fragmentation.

Male infertility has been associated with oxidative stress. Higher levels of reactive oxygen species (ROS) have been found in semen from men with low sperm count and motility, and poor sperm morphology, suggesting an imbalance in the redox system and an opportunity to use oxidative stress as a biomarker for semen quality. While several methods are available for measuring oxidative stress, they are not being implemented routinely in semen analysis likely because they are arduous and typically reflect only one side of the redox balance- oxidant activity.

A quick and all-inclusive measure of oxidative stress that could be used in a diagnostic setting (academic, hospital, clinical or reference laboratory) is the measure of static oxidation reduction potential (sORP) ; sORP reflects an integrated measure of the redox balance taking into account the activity of all oxidants (i.e. ROS, reactive nitrogen species, transition metal ions) and all antioxidants (i.e. small molecule antioxidants like ascorbate and enzymatic antioxidants like glutathione). Because sORP values are an integrated measures of both sides of the redox balance, sORP levels could be an identifying characteristic of semen quality.

The MiOXSYS System measures the redox balance by measuring sORP values. The MiOXSYS test results is used in conjunction with the established WHO semen analysis parameters. Previous studies suggest that increases in sORP are associated with lower sperm numbers, fewer motile sperm, and more abnormal sperm morphologies. The advantage of the MiOXSYS System is that sORP measures take into account both the oxidant and antioxidant sides of the redox balance, providing a rapid measure of oxidative stress, all with no sample preparation.

The objective of this study is to evaluate the performance of the MiOXSYS System as it measures sORP in semen samples with various degrees of semen quality. The MiOXSYS System is comprised of the MiOXSYS Analyzer and disposable, single-use MiOXSYS Sensors. Thirty microliters (30 uL) of neat semen is required for each test. sORP results from each semen sample will be compared to their corresponding results on the WHO semen analysis parameters (5th Edition Laboratory Manual for the Examination and Processing of Human Semen [2010]), which is the current methods for assessing semen quality.

ELIGIBILITY:
Inclusion Criteria:

1. Between 21 and 45 years of age, inclusive.
2. Male at birth.
3. Sexually abstinent for a minimum of 48 hours.
4. Sexually abstinent for no more than 7 days.
5. Provides written informed consent.
6. Agrees to complete all aspects of the study.

Exclusion Criteria:

1. Diagnosis of azoospermia.
2. Study participant on a previous date.
3. Unable to complete all aspects of the study.
4. Enrolled in another clinical study at the time of screening.
5. Diagnosed and/or is taking chronic medication for a chronic gastrointestinal condition including irritable bowel syndrome, colitis, or similar metabolic dietary conditions.
6. History of prostate cancer or any cancer that has been active over the last 5 years.
7. Vasectomy.
8. Surgery in the previous 90 days.
9. Trauma in the previous 90 days.
10. Takes additional daily antioxidant supplements including Vitamin C, Beta-Carotene, Vitamin E, Zinc, N-acetylcysteine, or Selenium. Multivitamin is acceptable for inclusion into the study.
11. Semen sample does not liquefy in 60 minutes.
12. White blood cells and/or round cells are greater than or equal to 1 million sperm/mL.
13. Sperm concentration in semen sample is less than 1 million sperm/mL.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Human males interested in fertility
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Static Oxidation Reduction Potential (sORP) between Normal and Abnormal semen samples | Semen samples, collected in accordance with published guidelines, will be tested within 1 hour of liquefaction
  Determine potential differences in sORP between the group of semen samples ("Normal") that meet WHO parameters for normal (good quality) semen and the group of semen samples ("Abnormal") that fail one or more WHO parameters (see Group description above). sORP is recorded as millivolts per sperm concentration (mV/million sperm/mL).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Miami, Miami, Florida
  - Tulane University, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Odessa Regional Medical Center, Odessa, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agarwal A, Sharma RK, Sharma R, Assidi M, Abuzenadah AM, Alshahrani S, Durairajanayagam D, Sabanegh E. Characterizing semen parameters and their association with reactive oxygen species in infertile men. Reprod Biol Endocrinol. 2014 May 7;12:33. doi: 10.1186/1477-7827-12-33. PMID 24885775
- [Background] Agarwal A, Mulgund A, Alshahrani S, Assidi M, Abuzenadah AM, Sharma R, Sabanegh E. Reactive oxygen species and sperm DNA damage in infertile men presenting with low level leukocytospermia. Reprod Biol Endocrinol. 2014 Dec 19;12:126. doi: 10.1186/1477-7827-12-126. PMID 25527074
- [Background] Du Plessis SS, Agarwal A, Halabi J, Tvrda E. Contemporary evidence on the physiological role of reactive oxygen species in human sperm function. J Assist Reprod Genet. 2015 Apr;32(4):509-20. doi: 10.1007/s10815-014-0425-7. Epub 2015 Feb 3. PMID 25646893
- [Background] Agarwal A, Sharma R, Roychoudhury S, Du Plessis S, Sabanegh E. MiOXSYS: a novel method of measuring oxidation reduction potential in semen and seminal plasma. Fertil Steril. 2016 Sep 1;106(3):566-573.e10. doi: 10.1016/j.fertnstert.2016.05.013. Epub 2016 May 31. PMID 27260688